CLINICAL TRIAL: NCT02146222
Title: Pharmacodynamic Study Using FLT-PET/CT in Patients With Advanced Solid Malignancies Treated With a Sequential Combination of X-82 and Docetaxel
Brief Title: VEGFR/PDGFR Dual Kinase Inhibitor X-82 and Docetaxel in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Tyrogenex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW13112; NCI-2014-00944 (Registry Identifier: NCI Trial ID); 2014-0528 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2014-05-20; First posted 2014-05-23 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2018-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Docetaxel; alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (high dose X-82, docetaxel) (Experimental): Patients receive high dose VEGFR/PDGFR dual kinase inhibitor X-82 PO QD on days 2-15. Beginning course 2, patients also receive docetaxel IV over 60 minutes on day 1.
  Interventions: Drug: VEGFR/PDGFR dual kinase inhibitor X-82; Drug: docetaxel; Other: fluorine F 18 fluorothymidine; Procedure: positron emission tomography/computed tomography; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (low dose X-82, docetaxel) (Experimental): Patients receive low dose VEGFR/PDGFR dual kinase inhibitor X-82 PO QD on days 2-15 and docetaxel IV as in Arm I.
  Interventions: Drug: VEGFR/PDGFR dual kinase inhibitor X-82; Drug: docetaxel; Other: fluorine F 18 fluorothymidine; Procedure: positron emission tomography/computed tomography; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: VEGFR/PDGFR dual kinase inhibitor X-82 — Given PO
  Other Names: X-82
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Other: fluorine F 18 fluorothymidine — Undergo FLT PET/CT
  Other Names: 18F-FLT; 3'-deoxy-3'-[18F]fluorothymidine; fluorothymidine F-18
Procedure: positron emission tomography/computed tomography — Undergo FLT PET/CT
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This partially randomized phase I trial studies the side effects and how well sequential dosing of vascular endothelial growth factor receptor (VEGFR)/platelet derived growth factor receptor (PDGFR) dual kinase inhibitor X-82 and docetaxel works in treating patients with solid tumors. VEGFR/PDGFR dual kinase inhibitor X-82 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving VEGFR/PDGFR dual kinase inhibitor X-82 and docetaxel one at a time instead of concurrently may work in treating patients with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of intermittent X-82 (VEGFR/PDGFR dual kinase inhibitor X-82) when administered in a 2 week on, 1 week off schedule (Cycle #1).

II. To evaluate the safety and tolerability of intermittent X-82 administered in combination with docetaxel every 3 weeks (Cycle #2).

III. To determine the change in vascular parameters using 3'Deoxy-3'-fluorothymidine (FLT) positron emission tomography (PET)/computed tomography (CT) to X-82 alone (Cycle #1).

IV. To determine the change in vascular parameters using FLT PET/CT to X-82 in combination with docetaxel (Cycle #2).

SECONDARY OBJECTIVES:

I. To determine the objective response using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 of intermittent X-82 with docetaxel.

II. To measure the change in plasma vascular endothelial growth factor (VEGF) levels with changes on FLT PET/CT.

III. To measure changes in X-82 pharmacokinetics with changes on FLT PET/CT.

TERTIARY OBJECTIVES:

I. To evaluate the safety and tolerability of sequential X-82 with docetaxel in disease sub-populations. (Dose expansion cohort) II. To evaluate the objective response rate of sequential X-82 with docetaxel in these disease sub-populations. (Dose expansion cohort)

OUTLINE: Patients are randomized to 1of 2 treatment arms.

ARM I: Patients receive high dose VEGFR/PDGFR dual kinase inhibitor X-82 orally (PO) once daily (QD) on days 2-15. Beginning course 2, patients also receive docetaxel intravenously (IV) over 60 minutes on day 1.

ARM II: Patients receive low dose VEGFR/PDGFR dual kinase inhibitor X-82 PO QD on days 2-15 and docetaxel IV as in Arm I.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

EXPANSION COHORT: Patients receive VEGFR/PDGFR dual kinase inhibitor X-82 as in Arm I and docetaxel IV over 60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* For the pharmacodynamic (PD) cohort, patients must have histologically or cytologically confirmed solid malignancy (excluding lymphoma) that is metastatic or unresectable; all patients will need to be approved by the principal investigator [PI] as certain diseases may not be appropriate for the imaging assessments)
* For the dose expansion cohort, patients with histologically or cytologically confirmed solid malignancy are eligible for treatment as long as insurance approval for docetaxel is obtained.
* Patients must have no available therapies that will confer clinical benefit and docetaxel is a reasonable treatment option for their malignancy
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 2 times the slice width with spiral CT scan (i.e. 10 mm if the CT slice width is 5 mm, 14 mm if the CT slice width is 7 mm)
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Serum calcium =< 12.0 mg/dL
* Total serum bilirubin =< institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine =< 1.5 mg/dL OR creatinine clearance (measured) >= 50 mL/min
* Urinary protein =< 2+ by urine analysis; if urine protein is > 2+ then a 24-hour urine collection can be done and the patient may enter only if urinary protein is < 2 g per 24 hours
* All patients need to be willing to undergo planned pharmacodynamic assessments, including serial PET imaging and pharmacokinetic sampling
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; all women of childbearing potential must have a negative pregnancy test prior to receiving X-82; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, experimental therapy or major surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered (to grade =< 1 or baseline) from clinically significant adverse events due to agents administered more than 4 weeks earlier (alopecia and fatigue excluded); clinical significance to be determined by investigator
* Patients may not be receiving any other investigational agents
* Prior anti-VEGF directed therapy may be allowed only if approved by the PI
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to X-82 or docetaxel
* Patients with poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher) are ineligible; patients with a history of hypertension (HTN) and stable blood pressure (BP) < 140/90 on anti-HTN regimen are eligible
* Patients will be required to have a baseline electrocardiogram (EKG) prior to the start of treatment; patients with a corrected QT (QTc) > 480 millisecond (ms) are excluded from the study
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain X-82 tablets are excluded
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 28 days of treatment
  * Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
  * History of myocardial infarction, ventricular arrhythmia, stable/unstable angina, symptomatic congestive heart failure, coronary/peripheral artery bypass graft or stenting or other significant cardiac disease within 12 months prior to study entry
  * Any history of arterial or venous thrombosis/thromboembolic event, including pulmonary embolism within the past 12 months
  * Any episode of atrial fibrillation in the prior 12 months
* Patients without appropriate lesion on CT scan for fluorothymidine (FLT)-PET/CT imaging will be excluded
* The eligibility of patients taking medications that are potent inducers or inhibitors of the cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) liver enzyme will be determined following a review of their case by the principal investigator; every effort should be made to switch patients taking such agents or substances to other medications; any identified agent needs to be stopped at least 2 weeks prior to study registration
* Patients with known brain metastases should be excluded; patients who had definitive treatment for their brain metastases which includes surgical resection/stereotactic body radiation therapy (SBRT) with whole brain radiation therapy (WBRT) > 6 months ago will be eligible
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infections or psychiatric illness/social situations that would limit compliance with study requirements are ineligible
* Pregnant women are excluded from this study; breastfeeding should be discontinued prior to starting study treatment
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients taking herbal supplements (St. John's Wort, gingko balboa, etc.) should discontinue these supplements two weeks prior to study registration
* Patients cannot be receiving concomitant chemotherapy, radiotherapy, experimental therapy or any other therapy for the purposes of anti-cancer treatment
* Subjects must not have clinically significant bleeding (i.e. GI bleed, intracranial bleeding) whtin 6 months or have had major surgery within 4 weeks. Minor surgeries (i.e. port placement, cataract surgery) are allowed if completed more than within 2 weeks from the start of treatment.
* Any brain metastases must be stable and not progressing prior to study entry
* Patients with prior malignancy except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated Stage I or II cancer from which the patient is currently in complete remission and has been disease free for the past 2 years
  * Any other cancer from which the patient has been disease-free for 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 (Pharmacodynamic study) | Up to 2 years
  The number and severity of toxicities and adverse events will be summarized using frequencies and percentages and stratified by X-82 dose level (low or high) and treatment (X-82 alone or X-82/docetaxel). Ninety-five percent confidence intervals for the toxicity rates will be constructed.
Changes in the FLT PET/CT vascular parameters for VEGF/PDGF dual kinase inhibitor X-82 | Baseline to day 15 (course 1)
  The changes in FLT PET/CT parameters will be calculated and summarized using descriptive statistics and compared using a paired t-test or non-parametric Wilcoxon signed rank test.
Changes in the FLT PET/CT vascular parameters for the combination of VEGFR/PDGFR dual kinase inhibitor X-82 and docetaxel | Day 1 to day 15 (course 2)
  The changes in FLT PET/CT parameters will be calculated and summarized using descriptive statistics and compared using a paired t-test or non-parametric Wilcoxon signed rank test.

SECONDARY OUTCOMES:
Disease response assessed by the RECIST 1.1 | Up to 2 years
  All patients with measurable disease will be classified as having either progressive disease (PD), stable disease (SD), a partial response (PR), or a complete response (CR). Responses will be summarized in tabular format delineating complete and partial responses as well as stable and progressive disease. A ninety-five percent confidence interval for the RECIST response rate will be constructed for the X-82 (low and high dose)/docetaxel combination.
Changes in VEGF | Baseline to up day 15 (course 2)
  Changes in VEGF levels will be summarized using descriptive statistics. Pearson's or Spearman's rank correlation analysis will be used to correlate changes in VEGF and pharmacokinetic parameters with changes in FLT PET/CT parameters.
Pharmacokinetic parameters of VEGFR/PDGFR dual kinase inhibitor X-82 | Within 3 hours prior to X-82 administration on days 1, 12-15, and 19-21 (course 1); and days 12-15 (course 2)
  Changes in X-82 pharmacokinetics will be summarized using descriptive statistics. Pearson's or Spearman's rank correlation analysis will be used to correlate changes in VEGF and pharmacokinetic parameters with changes in FLT PET/CT parameters.

OTHER OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The objective response rate will be summarized in tabular format delineating CR and PR as well as SD and PD. The posterior distributions of the ORR for each disease cohort will be computed using the Gibbs sampling algorithm, based on a Bayesian hierarchical model. Summaries of the posterior distribution including the mean, median and variance along with 95% credible intervals will be provided for each disease cohort and for all cohorts combined.
Incidence of toxicity graded according to NCI CTCAE version 4.0 (Dose expansion study) | Up to 2 years
  The number and severity of toxicities and adverse events will be summarized using frequencies and percentages and stratified by disease cohort. Ninety-five percent confidence intervals for the toxicity rates will be constructed.

CONTACTS AND LOCATIONS:
Overall Officials: Justine Bruce, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Jackson TL, Boyer D, Brown DM, Chaudhry N, Elman M, Liang C, O'Shaughnessy D, Parsons EC, Patel S, Slakter JS, Rosenfeld PJ. Oral Tyrosine Kinase Inhibitor for Neovascular Age-Related Macular Degeneration: A Phase 1 Dose-Escalation Study. JAMA Ophthalmol. 2017 Jul 1;135(7):761-767. doi: 10.1001/jamaophthalmol.2017.1571. PMID 28570723
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/